CLINICAL TRIAL: NCT02842736
Title: A CLinical Study to Evaluate the Safety And Effectiveness of the CeRene DevIce to Treat HeavY Menstrual Bleeding
Acronym: CLARITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Channel Medsystems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0101
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Menorrhagia
Keywords: heavy menstrual bleeding; endometrial ablation
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Endometrial Cryoablation (Experimental)
  Interventions: Device: Cerene(R) Cryotherapy Device

INTERVENTIONS:
Device: Cerene(R) Cryotherapy Device

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the Cerene Cryotherapy Device in reducing menstrual bleeding in women with heavy menstrual bleeding (menorrhagia) due to benign causes for whom child bearing is complete.

ELIGIBILITY:
Inclusion Criteria:

* Refractory heavy menstrual bleeding with no definable organic cause
* Female subject age 25 to 50 years, inclusive
* Sounded length of uterine cavity no greater than 10 cm and endometrial cavity no greater than 6.5 cm
* Sufficient myometrial thickness
* Documented excessive menstrual blood loss within 3 months of informed consent
* Premenopausal confirmed by follicle stimulating hormone (FSH) measurement
* Agrees to use a reliable form of contraception following ablation treatment
* Provides written informed consent using a form that has been approved by the reviewing ethics committee
* Agrees to follow-up exams and data collection requirements
* Demonstrates an understanding of how to record menstrual blood loss using a menstrual pictogram
* Has predictable, cyclic menstrual cycles

Exclusion Criteria:

* Pregnant or has a desire to conceive
* Endometrial hyperplasia as confirmed by histology
* Active endometritis
* Active pelvic inflammatory disease
* Active sexually transmitted disease (STD)
* Presence of bacteremia, sepsis, or other active systemic infection
* Active infection of the genitals, vagina, cervix, or uterus
* Known/suspected abdominal, pelvic, or gynecological malignancy within the past 5 years
* Known clotting defects or bleeding disorders
* Abnormal cytology on Human papillomavirus (HPV) testing not treated according to local standards.
* Prior uterine surgery that interrupts the integrity of the uterine wall (e.g., transmural myomectomy or classical cesarean section).
* Previous low transverse cesarean section where the myometrial wall thickness is insufficient
* Previous endometrial ablation procedure
* Clinically significant adenomyosis indicated by subject complaints, imaging, or clinician's judgment
* Presence of an implantable contraceptive device
* Currently on medications that could thin the myometrial muscle
* Currently on anticoagulants
* Abnormal or obstructed cavity
* Currently using an intrauterine device (IUD) and unwilling to remove the IUD
* Post-partum ≤ 6-months
* Considering participation in a research study of an investigational drug or device that would begin during the course of this investigational study
* Any general health or mental, or other situation or condition which, in the opinion of the Investigator, could represent an increased risk for the subject or impact the subject's ability to comply with protocol requirements

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - WomanCare PC, Arlington Heights, Illinois
  - The Advance Gynecologic Surgery Institute, Naperville, Illinois
  - Women's Health Advantage, Fort Wayne, Indiana
  - Basinski LLC, Newburgh, Indiana
  - Asheville Women's Medical Center, Asheville, North Carolina
  - Seven Hills Women's Health, Cincinnati, Ohio
  - Amy Brenner MD and Associates, LLC, Mason, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Premier Clinical Research, Spokane, Washington
- Canada (2):
  - Allan Centre, Calgary, Alberta
  - LaSalle Hospital, LaSalle, Quebec
- Hospital Universitario de la Universidad Autónoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Derived] Curlin HL, Anderson TL. Endometrial Cryoablation for the Treatment of Heavy Menstrual Bleeding: 36-Month Outcomes from the CLARITY Study. Int J Womens Health. 2022 Aug 10;14:1083-1092. doi: 10.2147/IJWH.S371044. eCollection 2022. PMID 35983177
- [Derived] Curlin H, Cholkeri-Singh A, Leal JGG, Anderson T. Hysteroscopic Access and Uterine Cavity Evaluation 12 Months after Endometrial Ablation with the Cerene Cryotherapy Device. J Minim Invasive Gynecol. 2022 Mar;29(3):440-447. doi: 10.1016/j.jmig.2021.11.016. Epub 2021 Nov 25. PMID 34839060
- [Derived] Curlin HL, Cintron LC, Anderson TL. A Prospective, Multicenter, Clinical Trial Evaluating the Safety and Effectiveness of the Cerene Device to Treat Heavy Menstrual Bleeding. J Minim Invasive Gynecol. 2021 Apr;28(4):899-908. doi: 10.1016/j.jmig.2020.08.013. Epub 2020 Aug 22. PMID 32835865

RESULTS

PARTICIPANT FLOW:
Groups:
- Endometrial Cryoablation: Cerene(R) Cryotherapy Device
Period: Overall Study
Arm/Group | Endometrial Cryoablation
Started | 242 (Treated)
Known Month 12 Outcome | 230
24 Month Visit Performed | 210
Completed | 201 (36 Month Visit Completed)
Not Completed | 41
Not completed — Lost to Follow-up | 13
Not completed — Intervention for menstrual bleeding | 17
Not completed — Withdrawal by Subject | 4
Not completed — Pregnancy | 3
Not completed — Hysterectomy for fibroids | 2
Not completed — Hysterectomy for uterine prolapse | 1
Not completed — IUD: Mirena | 1

BASELINE CHARACTERISTICS:
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 190
  Black or African American | 6
  American Indian or Alaska Native | 3
  Other | 43
Baseline PBLAC (Pictorial Blood Loss Assessment Chart) Score [Mean (Standard Deviation); unit: scores on a scale] — Scale information for PBLAC (Pictorial Blood Loss Assessment Chart):
  The scale minimum is 0, which indicates amenorrhea, i.e. no bleeding. There is no scale maximum. A score of 100 indicates eumenorrhea, i.e. normal menstrual bleeding. A lower PBLAC score indicates less bleeding; a higher PBLAC score indicates more bleeding.
  At baseline, the range of PBLAC values was 150.0 to 4506.5.
  scores on a scale | 360.6 (332.1)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Number of Serious Adverse Events and Serious Device-related Adverse Events
Time Frame: 12 months
Population: The Intent-to-Treat (ITT) population is comprised of all patients who successfully completed screening and presented on the day of treatment.
Measure: Number; unit: Reports of events
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 242
Reports of events
  Serious adverse events | 7
  Serious device-related adverse events | 0

2. Primary Outcome: Primary Effectiveness Endpoint: Number of Subjects With Reduction in Menstrual Bleeding to PBLAC Score of ≤75
Description: Success for the primary effectiveness endpoint was defined as reduction in menstrual bleeding to a PBLAC (Pictorial Blood Loss Assessment Chart) score of ≤75.
  Scale information for PBLAC (Pictorial Blood Loss Assessment Chart):
  The scale minimum is 0, which indicates amenorrhea, i.e. no bleeding. There is no scale maximum. A score of 100 indicates eumenorrhea, i.e. normal menstrual bleeding. A lower PBLAC score indicates less bleeding; a higher PBLAC score indicates more bleeding.
Time Frame: 12 months
Population: The Intent-to-Treat (ITT) population comprised all patients who successfully completed screening and presented on the day of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 242
Participants | 186

3. Secondary Outcome: Dysmennorhea
Description: Subjects were queried regarding if they suffer from dysmenorrhea (painful cramping associated with menstruation). The subject was asked to rate their level of dysmenorrhea on a scale from 0 to 5, with 0 indicating no symptoms and 5 indicating very severe symptoms. A score of 0 was considered better than a score of 5.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 230
Participants
  0 - No symptom | 74
  1 - Very Mild | 70
  2 - Mild | 40
  3 - Moderate | 33
  4 - Severe | 10
  5 - Very Severe | 3

4. Secondary Outcome: Amenorrhea
Description: Pictorial blood loss assessment (PBLAC) score = 0
  Scale information for PBLAC (Pictorial Blood Loss Assessment Chart):
  The scale minimum is 0, which indicates amenorrhea, i.e. no bleeding. There is no scale maximum. A score of 100 indicates eumenorrhea, i.e. normal menstrual bleeding. A lower PBLAC score indicates less bleeding; a higher PBLAC score indicates more bleeding.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 242
Participants | 25

5. Secondary Outcome: Investigator Evaluation of the Uterine Cavity
Time Frame: 12 Months
Population: Of 230 subjects with a known Month 12 outcome, 223 underwent a hysteroscopy at Month 12. The remaining seven (7) subjects encountered scheduling conflicts or illness.
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 223
Participants
  Uterine cavity entry with a hysteroscope: YES | 220
  Uterine cavity entry with a hysteroscope: NO | 3
  Full visualization of the uterine cavity: YES | 204
  Full visualization of the uterine cavity: NO | 19

6. Secondary Outcome: Investigator Assessment of Cavity Findings
Description: Questions to the investigator
Time Frame: 12 Months
Population: Investigators' assessment was based on the 204 subjects whose cavities could be fully visualized (see Secondary Outcome: Investigator Evaluation of the Uterine Cavity).
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 204
Participants
  Would the Investigator be able to direct a biopsy anywhere within the uterine cavity?: YES | 178
  Would the Investigator be able to direct a biopsy anywhere within the uterine cavity?: NO | 26
  Satisfied with ability to adequately visualize the endometrium to evaluate for pathologic change?: YES | 195
  Satisfied with ability to adequately visualize the endometrium to evaluate for pathologic change?: NO | 9

7. Secondary Outcome: Anesthesia and Pain Medications at Treatment
Time Frame: Day of Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 242
Participants
  Paracervical block only | 20
  Paracervical block with nonsteroidal anti-inflammatories | 48
  Paracervical block with oral narcotics and/or anxiolytics | 167
  Paracervical block with intravenous sedation | 7
  General anesthesia | 0

8. Secondary Outcome: Subject Rating of Pain During Treatment and Day One Post-Treatment
Description: Pain rating using numeric rating scale, minimum 0, maximum 10, with 0 designated as no pain and 10 designated as the worst pain.
Time Frame: Day of Treatment and Day One Post-Treatment
Population: Some subjects did not provide a pain score rating due to sedation. One subject did not provide a pain score at her Day 1 visit.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 242
units on a scale
  Before Device Insertion: number analyzed (Participants) | 241
  Before Device Insertion | 1 [0 to 10]
  After Device Insertion: number analyzed (Participants) | 240
  After Device Insertion | 2 [0 to 10]
  After Liner Deployment (before endometrial ablation was initiated): number analyzed (Participants) | 240
  After Liner Deployment (before endometrial ablation was initiated) | 1 [0 to 10]
  After 1 Minute of Ablation: number analyzed (Participants) | 240
  After 1 Minute of Ablation | 2 [0 to 10]
  End of Ablation: number analyzed (Participants) | 239
  End of Ablation | 1 [0 to 10]
  15-30 Minutes Post-Procedure | 2 [0 to 10]
  At Time of Discharge | 2 [0 to 8]
  Day 1: number analyzed (Participants) | 241
  Day 1 | 0 [0 to 8]

9. Other Pre Specified Outcome: Subjects' Report of Their Last Menstrual Period
Description: Subjects were asked to describe their last menstrual period
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 201
Participants
  I no longer get my period | 29
  My periods are lighter than normal | 99
  My periods are normal | 50
  I continue to have heavy periods | 23

10. Other Pre Specified Outcome: Menstrual Impact Questionnaire
Description: Subjects' Report of Activity Limitations
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 201
Participants
  Free of limitation in activity at moderate or higher level | 182
  Limitation in activity is present at moderate or higher level | 19

11. Other Pre Specified Outcome: Premenstrual Symptoms Impact Survey
Description: Subjects' Report of Pre-Menstrual Symptoms (PMS)
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 201
Participants
  Free of PMS often, most often, very often, or all of the time | 171
  PMS occur often, most often, very often, or all of the time | 30

12. Other Pre Specified Outcome: Subject Satisfaction
Description: Subject's level of satisfaction with the results of her Cerene treatment
Time Frame: 36 Months
Population: Of 201 subjects who completed the study, 181 reported their level of satisfaction
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 181
Participants
  Satisfied or very satisfied | 153
  Dissatisfied or very dissatisfied | 28

13. Other Pre Specified Outcome: Subject Recommendation
Description: Subjects' reported level of recommendation to a friend/family
Time Frame: 36 months
Population: Of 201 subjects who completed the study, 193 reported their level of recommendation
Measure: Count of Participants; unit: Participants
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 193
Participants
  Definitely or maybe recommend | 175
  Probably not or definitely not recommend | 18

14. Other Pre Specified Outcome: Procedure Time
Description: Device insertion to device removal
Time Frame: Day of Treatment
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 242
minutes | 6.9 (1.1)

15. Other Pre Specified Outcome: Return to Normal Daily Activities
Time Frame: Two-Weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Endometrial Cryoablation
Number analyzed (Participants) | 242
days | 2.0 (2.3)

ADVERSE EVENTS:
Time Frame: 36 Months
Description: Adverse event information was collected throughout the study at each subject contact. All serious adverse events observed in the study are reported in "Serious Adverse Events" below. "Other (Not Including Serious) Adverse Events" below presents a summary of (1) for up to 12-month follow-up, device and/or procedure-related non-serious adverse events occurring in more than 1% of subjects and (2) for post 12-Month follow-up, all gynecologic adverse events.
Arm/Group | Endometrial Cryoablation
All-Cause Mortality (participants affected / at risk) | 0/242
Serious Adverse Events (participants affected / at risk) | 6/242
Other Adverse Events (participants affected / at risk) | 29/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometrial Cryoablation (N=242)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Acute Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bile Duct Obstruction (Hepatobiliary disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Chronic Constipation (Gastrointestinal disorders) | 1 (1)
Paresthesia of limbs (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endometrial Cryoablation (N=242)
Bacterial vaginosis (Infections and infestations) | 7 (7)
Presyncope (Nervous system disorders) | 3 (4)
Uterine cramps (Reproductive system and breast disorders) | 8 (8)
Emesis (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Endometritis (Infections and infestations) | 1 (1)
Vulvovaginitis Streptococcal (Infections and infestations) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Menstrual cramps (Reproductive system and breast disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Uterine tenderness (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) — Gynecologic adverse event reported after Month 12
Dysmenorrhea (Reproductive system and breast disorders) | 2 (2) — Gynecologic adverse event reported after Month 12
Dyspareunia (Reproductive system and breast disorders) | 1 (1) — Gynecologic adverse event reported after Month 12
Endometritis (Reproductive system and breast disorders) | 1 (1) — Gynecologic adverse event reported after Month 12
Intermenstrual bleeding (Reproductive system and breast disorders) | 2 (2) — Gynecologic adverse event reported after Month 12
Menorrhagia (Reproductive system and breast disorders) | 15 (15) — Gynecologic adverse event reported after Month 12
Pelvic cramping (Reproductive system and breast disorders) | 2 (2) — Gynecologic adverse event reported after Month 12
Pelvic pain (Reproductive system and breast disorders) | 4 (4) — Gynecologic adverse event reported after Month 12
Polycystic ovarian disease (Reproductive system and breast disorders) | 1 (1) — Gynecologic adverse event reported after Month 12
Pos- coital bleeding (Reproductive system and breast disorders) | 1 (1) — Gynecologic adverse event reported after Month 12
Pregnancy; uterine (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Gynecologic adverse event reported after Month 12
Pregnancy; uterine terminated (Pregnancy, puerperium and perinatal conditions) | 1 (1) — Gynecologic adverse event reported after Month 12
Right breast mass (Reproductive system and breast disorders) | 1 (1) — Gynecologic adverse event reported after Month 12
Uterine fibroids (Reproductive system and breast disorders) | 2 (2) — Gynecologic adverse event reported after Month 12
Uterine prolapse Stage 2 (Reproductive system and breast disorders) | 1 (1) — Gynecologic adverse event reported after Month 12
Vaginal infection and/or discharge (Reproductive system and breast disorders) | 11 (11) — Gynecologic adverse event reported after Month 12
Vaginal/vulvar pruritus (Reproductive system and breast disorders) | 2 (2) — Gynecologic adverse event reported after Month 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators have the right to publish their data, with the following provisions: (1) investigators at academic centers have a time frame for submission of their manuscript, or other, to Sponsor prior to publication and (2) investigators at private clinics can request prior written consent.

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT02842736/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT02842736/SAP_001.pdf